CLINICAL TRIAL: NCT03702907
Title: DC Longitudinal Study on Aging and Specimen Bank
Acronym: (DC LSOA)
Status: Recruiting | Type: Observational
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, R. Scott Turner, Director, Georgetown University
Other Study IDs: 2007-249
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer Disease; Dementia; Mild Cognitive Impairment; Aging; Aging Disorder
Keywords: Frontotemporal Dementia; Lewy Body Dementia; Aging; Vascular Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Frontotemporal Dementia; Lewy Body Disease; Dementia, Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of Blood Collection of Cerebrospinal Fluid (CSF) (Optional)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Cognition: No diagnosis of a cognitive disorder
- Cognitive Disorder: Diagnosed with a cognitive disorder such as :Mild Cognitive Impairment, Alzheimer's disease, Frontotemporal Dementia, Lewy Body Dementia, Vascular Dementia, or other neurodegenerative condition.

SUMMARY:
The Georgetown University Memory Disorders Program, part of the Department of Neurology, is conducting pilot studies of the feasibility of various diagnostic tests for Alzheimer's disease, mild cognitive impairment and other neurodegenerative diseases. Further, this study is assessing longitudinal changes in biological, lifestyle, and cognitive assessment collection.

The primary goal of this study is to examine the feasibility of biochemical assays, genetic testing, and cognitive and lifestyle assessments in the ante-mortem diagnosis of Alzheimer's disease, mild cognitive impairment and other neurodegenerative diseases. This research involves genetic and cognitive status testing but the findings will not be shared with research subjects. This will be accomplished ex vivo using blood, and/or cerebrospinal fluid (CSF) specimens from patients with a diagnosis of probable Alzheimer's disease, mild cognitive impairment, or other neurodegenerative diseases and from normal controls.

DETAILED DESCRIPTION:
These studies will examine the feasibility of using various biochemical assays in blood, and/or cerebrospinal fluid, genetic testing, cognitive status assessments, and lifestyle questionnaires to aid in the ante-mortem diagnosis of Alzheimer's and other neurodegenerative diseases.

Subjects have 2 options for participation. They may solely participate in the main study or the main study and the longitudinal substudy. The main study includes a single visit at which demographic and medical information will be recorded, brief cognitive testing, and blood and/or cerebrospinal fluid (CSF)(optional) specimens will be collected for the research assays. Genetic testing will take place. No clinical laboratory testing will be done and no results will be communicated to subjects.

During the Longitudinal substudy, each subject will be asked to participate in ongoing longitudinal study visits at which demographic and medical information will be recorded, cognitive testing and lifestyle questionnaire collection will occur, and blood and/or cerebrospinal fluid (CSF) specimens will be collected for the research assays. I

If one is eligible and agrees to participate in the longitudinal sub-study, they will be asked to come into the clinic for an Initial Study Visit, and then return every year or every other year, depending on which group they fit into (Cognitively Normal (CN), Mild Cognitive Impairment (MCI), Alzheimer's Disease (AD), other neurodegenerative disease) for ongoing Follow-Up Clinic Visits.

CN participants will come into the clinic every other year, with telephone checks occurring on alternating years, until the study ends.

MCI, AD, and other participants with a diagnosis of any other neurodegenerative disease will come into the clinic every year until the study ends.

Those in the Cognitively Normal group, will also partake in a short Telephone Visit on the year that they do not come into the clinic. This phone call will be done only to assess/update your medical history and medications.

Genetic testing will take place. No clinical laboratory testing will be done and no results will be communicated to subjects. Those who are deemed to be cognitively normal, assessed by cognitive status instruments, will be asked to return to the clinic for ongoing study visits every other year, with telephone visits on the off year. Those who have a diagnosis of MCI, AD, or any other neurodegenerative disease will be asked to return to the clinic yearly for their longitudinal follow-up study visits.

For both the main and longitudinal sub-study, specimens will be banked for future use and can be provided to other researchers at Georgetown University, other institutions or commercial enterprise in a de-identified manner through a formal request system. For all investigators, not affiliated with the Memory Disorders Program, a formal request will be submitted to the PI for review. If the request is approved, requested specimens and/or data from the study will be sent in a de-identified manner to ensure date security and privacy. The reason for the option of data sharing is to enhance exploration of different lines of analysis, and assist emerging investigators with access to a database with robust data and specimen collections.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 and older.
* Subjects within the age range of 45-50 years old must have a first degree relative with a neurodegenerative disease.

Exclusion Criteria:

* Individuals under 45 years of age

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All genders, races, and ethnicities eligible. Normal controls and those diagnosed with a neurodegenerative disorder eligible.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
CDR | 9 years
  Clinical Dementia Rating

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Memory Disorders Program, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Program Website — https://memory.georgetown.edu/